CLINICAL TRIAL: NCT05542095
Title: Simvastatin Nasal Rinses for the Treatment of COVID-19 Mediated Dysomsia
Acronym: SimCA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely; IRB approval not obtained
Sponsor: Washington University School of Medicine (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Nyssa Farrell, Assistant Professor of Otolaryngology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SimCA Trial
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Olfactory Disorder; COVID-19
Keywords: Olfactory Disorder; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: This is an open-label phase 1 trial of topical simvastatin delivered via nasal irrigation using a standard three plus three (3+3) dose-escalation design. Subjects are entered into the study in groups of 3. The study will continue with successive cohorts of 3 subjects until dose-limiting toxicities (DLT) are observed in greater than 33% of the enrolled subjects. DLT is defined as the development of statin intolerance with liver toxicity or muscle toxicity or the development of significant systemic or sinonasal symptoms requiring drug discontinuation. The first cohort will receive the lowest dose of simvastatin (0.1mg) via nasal irrigation for 4 weeks. The next group of 3 subjects will receive the consecutive higher dose of simvastatin. We anticipate that 4 doses will be trialed (0.1 mg, 0.25 mg, 0.5 mg, 1 mg) within the predetermined safety range.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- topical nasal simvastatin - 0.1 mg dose (Experimental): topical nasal simvastatin - 0.1 mg dose
  Subjects are entered into the study in groups of 3. This first cohort will receive the lowest dose of simvastatin (0.1mg) via nasal irrigation for 4 weeks. If none of the 3 subjects report toxicity, the next group of 3 subjects enrolled will receive the consecutive higher dose of simvastatin for 1 month. If >2 of the 3 subjects enrolled in the first group report toxicity then the dose is considered toxic or "MTD is exceeded." If 1 of the first 3 reports toxicity, then the next group of 3 enrolled subjects will receive the same dose as group 1. When 6 subjects receive the same dose, and <1 of them report toxicity, the consecutive group of 3 subjects will receive the successive higher dose. If >2 of the 6 subjects on the same dose report toxicities, then MTD is exceeded. Intra-patient dose escalation will not be performed.
  Interventions: Drug: Simvastatin
- topical nasal simvastatin - 0.25 mg dose (Experimental): topical nasal simvastatin - 0.25 mg dose
  Subjects are entered into the study in groups of 3. This 2nd cohort will receive the 0.25mg simvastatin via nasal irrigation for 4 weeks. If none of the 3 subjects report toxicity, the next group of 3 subjects enrolled will receive the consecutive higher dose of simvastatin for 1 month. If >2 of the 3 subjects enrolled in the first group report toxicity then the dose is considered toxic or "MTD is exceeded." If 1 of the first 3 reports toxicity, then the next group of 3 enrolled subjects will receive the same dose as group 1. When 6 subjects receive the same dose, and <1 of them report toxicity, the consecutive group of 3 subjects will receive the successive higher dose. If >2 of the 6 subjects on the same dose report toxicities, then MTD is exceeded. Intra-patient dose escalation will not be performed.
  Interventions: Drug: Simvastatin
- topical nasal simvastatin - 0.5 mg dose (Experimental): topical nasal simvastatin - 0.5 mg dose
  Subjects are entered into the study in groups of 3. This 3rd cohort will receive the 0.5mg simvastatin via nasal irrigation for 4 weeks. If none of the 3 subjects report toxicity, the next group of 3 subjects enrolled will receive the consecutive higher dose of simvastatin for 1 month. If >2 of the 3 subjects enrolled in the first group report toxicity then the dose is considered toxic or "MTD is exceeded." If 1 of the first 3 reports toxicity, then the next group of 3 enrolled subjects will receive the same dose as group 1. When 6 subjects receive the same dose, and <1 of them report toxicity, the consecutive group of 3 subjects will receive the successive higher dose. If >2 of the 6 subjects on the same dose report toxicities, then MTD is exceeded. Intra-patient dose escalation will not be performed.
  Interventions: Drug: Simvastatin
- topical nasal simvastatin - 1 mg dose (Experimental): topical nasal simvastatin - 1 mg dose
  Subjects are entered into the study in groups of 3. This 4th cohort will receive the 1mg simvastatin via nasal irrigation for 4 weeks. If none of the 3 subjects report toxicity, then the drug will be considered tolerated at the maximum tested dose. If >2 of the 3 subjects enrolled in the first group report toxicity then the dose is considered toxic or "MTD is exceeded." If 1 of the first 3 reports toxicity, then the next group of 3 enrolled subjects will receive the same dose as group 1. When 6 subjects receive the same dose, and <1 of them report toxicity, then this maximum dose is considered tolerable. If >2 of the 6 subjects on the same dose report toxicities, then MTD is exceeded. Intra-patient dose escalation will not be performed.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Compounded simvastatin that is suspended within a nasal saline irrigation will be utilized throughout this study. Participants will suspend the contents of the simvastatin capsules (0.1mg, 0.25 mg, 0.5 mg, and 1 mg) into the sinus rinse bottle containing nasal saline. All participants will receive an 8-ounce sinus rinse bottle and a 4-week supply of USP Grade Sodium Chloride & Sodium Bicarbonate Mixture (pH balanced, Isotonic & Preservative & Iodine Free) commercially prepared packets. Participants will either need to purchase distilled water or boil tap water for five minutes for use with the saline irrigation.
  Other Names: ZOCOR

SUMMARY:
Olfactory dysfunction (OD) or changes in smell and/or taste is one of the cardinal presenting symptoms of COVID-19. Despite the prevalence of COVID and resultant OD, the pathophysiology of COVID-mediated OD is not fully understood, but recent evidence indicates that local inflammatory and oxidative injury play a major role.

This phase 1 safety trial evaluates the use of simvastatin nasal irrigations for the management of COVID-mediated OD. We will determine the maximum tolerable dose and evaluate the safety and tolerability of high-volume simvastatin nasal irrigations in subjects with persistent COVID-mediated OD.

Each subject will complete bloodwork at baseline and then at the completion of their participation in the study. During this trial, we will observe olfactory function for each participant at baseline and completion of this study via the University of Pennsylvania Smell Identification Test (UPSIT). Investigational product will be shipped directly to the subject for daily irrigation each day for 4 weeks. Weekly throughout the study for a total of 4 weeks, subjects will complete the Sino-Nasal Outcome Test-22.

The current study would provide the support for Phase II and III clinical trials. Additionally, the study has applications for other disease processes affecting the sinonasal cavities.

DETAILED DESCRIPTION:
Olfactory dysfunction (OD) is one of the hallmark symptoms of SARS-CoV-2, the virus which has caused the COVID-19 pandemic. There is increasing evidence of the role of local inflammation and oxidative damage in COVID-mediated OD. To date, the only recommended therapy for patients with COVID-19 mediated OD is olfactory training, which has not been shown to result in a dramatic improvement in olfaction. Thus, it is essential that other effective management strategies are identified for the rapidly growing COVID-mediated dysosmic population.

Statins are utilized primarily for the reduction of cholesterol. However, statins also have pleiotropic effects on cellular inflammation, oxidative stress, and neuroprotection. Multiple studies have evaluated the anti-inflammatory effects of topical statins within the airway and shown that topical application can reduce inflammatory mediators such as IL-4, IL-6, IL-6, IL-8, CCL-11 and inflammatory cells. The anti-inflammatory effect of statins has also been demonstrated for neuroinflammation. One study evaluated the anti-inflammatory effects of 10 uM simvastatin suspensions on human monocyte-derived macrophages THP-1 as a surrogate for microglial cells and noted a significant reduction in lipopolysaccharide-induced IL-6 secretion. Another study evaluated the impact of nasally administered polymerosomes impregnated with simvastatin (doses 0-20 ug/mL) and brain-derived neurotrophic factor on neuroinflammation in mice and noted reduced IL-6 and IL-1b within brain homogenate after 3 days of exposure.

The safety of topical simvastatin has also been explored in vitro. The effect of topical simvastatin on nasal ciliary function was evaluated by applying 1x10-6 M to nasal cell brushings for 30 minutes. The resulting ciliary beat frequency was evaluated and demonstrated no adverse effects compared to control. Transepithelial electrical resistance was also evaluated 4 hours after exposure of bronchial epithelial cells aerosolized simvastatin and did not demonstrate any significant changes in transepithelial cell resistance between control cells and those treated with aerosolized simvastatin short term. However, after 14 days, a significant reduction in transepithelial resistance was noted, indicating a significant increase in cellular permeability. It is important to note, however, that this change incellular permeability did not associate with any change in cell viability. Manickavasagam et al. also evaluated the safety of simvastatin nanoparticles up to 20 uM on mouse hippocampal neuronal cells and did not note toxicity, indicating that our test concentration (maximum 10 uM) should not result in toxicity to the neural tissue.

Wang et al. evaluated the toxicity and anti-inflammatory effects of statin suspensions applied to human nasal epithelial cells and showed a reduction in CCL5, CCL11, IL-5, and IL-13 after 24 hr drug exposure without significant impacts of cell viability.

Statins also aid in nerve regeneration. Multiple studies have demonstrated neuroprotective effects after spinal cord injury, traumatic brain injury, and peripheral nerve injury. Studies of peripheral nerve injury have demonstrated that early administration of statins can accelerate nerve regeneration through increased neurite growth. Multiple mouse studies have shown that oral statin administration can improve proliferation and neuroregenesis of the olfactory epithelium in mice who have undergone chemical injury to the olfactory mucosa.

Statins can likely safely treat COVID-mediated OD through their anti-inflammatory, anti-oxidant, and neuroregenerative capabilities. However, oral statin administration has very low bioavailability due to metabolism within the intestinal wall and high first-pass metabolism by the liver. Orally dosed statins also have a risk of statin intolerance, in which patients develop statin-associated muscle symptoms, ranging from mild myalgias to life-threatening rhabdomyolysis. As such, the administration of statins via non-oral routes could increase local bioavailability, improve drug efficacy, and allow for lower systemic doses, limiting the risk of adverse effects.

Intranasal drug administration through nasal irrigation has been widely used for the management of sinonasal disorders. There are many advantages of intranasal medications, including delivery of higher concentrations than by systemic routes, increased bioavailability by bypassing first-pass liver metabolism, rapid drug absorption and onset of action, reduced side effects, and the potential for direct nervous system absorption via the olfactory neuroepithelium. The nasal cavity presents multiple barriers to drug application: mucous layer, epithelial lining, and tight junctions. So, lipophilicity of a drug provides a major advantage, allowing the drug to penetrate the mucous layer and passively diffuse through the nasal epithelial cells.

Simvastatin, a highly lipophilic pro-drug, is ideal for nasal use. It is converted to its active hydrophilic form (simvastatin hydroxyacid) by cytochrome p450 enzyme 3A4/5, which is present within the nasal epithelium. Of the available statins, simvastatin has been frequently evaluated for its anti-inflammatory components in the lower airway. Many animal models have also demonstrated improved recovery of injured peripheral nerves after simvastatin administration. Topical simvastatin, with its high lipophilicity and pleiotropic effects on inflammation, oxidative stress, and neuroregenerative capacity make it the ideal statin for the topical application and management of COVID-mediated OD.

Our lab has performed evaluations of 0.1-10 mg custom compounded simvastatin suspended within 240 mL phosphate buffered saline (1-100 uM simvastatin). These suspensions were applied daily to the surface hTEC (differentiated at an air-liquid interface) for 5 min a day, followed by 2 saline rinses for a total of 4 days. The ciliary beat frequency (CBF), transepithelial resistance (TEER), and lactate dehydrogenase (LDH) were evaluated at time 0 and after 4 days of drug exposure. Cells were immunostained for cilia using an antibody to acetylated alpha tubulin and cell junctions using an antibody to E-cadherin. We found that cilia of multiciliated cells treated with simvastatin at 0.1-10 mg doses were not different from control. Similarly, E-cadherin was maintained except at the higher 5 mg dose. For cells treated with 0.1-1mg, there was no change in TEER after 4 days of drug exposure. However, a decrease was noted in TEER for cells treated with 5 and 10 mg simvastatin. Though TEER did decrease, there was no evidence of elevated LDH after 4 days of 0.1-10mg drug exposure, indicating that there was no cellular toxicity.

Given these findings, as well as previous data demonstrating anti-inflammatory effects of 10 uM (1 mg simvastatin within 240 mL saline) simvastatin suspensions, we propose a Phase 1 trial to analyze the safety and tolerability, as well as the maximum tolerable dose, of topical simvastatin nasal rinses in adults with COVID-mediated OD. The first cohort will receive the lowest dose of simvastatin (0.1 mg) via nasal irrigation for 4 weeks. If none of the 3 subjects report toxicity, the next group of 3 subjects enrolled will receive the consecutive higher dose of simvastatin for 1 month to a maximum dose of (1mg). We plan to test the following doses: 0.1 mg, 0.25 mg, 0.5 mg, 1 mg.

This is an open-label phase 1 trial of topical simvastatin delivered via nasal irrigation, which will be performed at a single tertiary academic medical center. We propose to use a standard three plus three (3+3) dose-escalation design. Investigational product will be shipped directly to the subject for daily irrigation each day for 4 weeks.

For subjects who meet inclusion criteria, the subject name, address, phone number, age, sex, and date/time of clinic visits related to OD will be obtained from the chart. The following baseline laboratory tests will be obtained prior to initiation of the trial to ensure that subjects do not have conditions that would increase the risk of statin intolerance: thyroid stimulating hormone (TSH), aspartate transaminase (AST), alanine transaminase (ALT), estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), creatinine (Cr), creatine kinase (CK), and total cholesterol. Subjects with lab values outside of the standard normal ranges will be excluded from the study and referred to their primary care physician (PCP). Prior to statin administration, all subjects will have an evaluation with rigid nasal endoscopy by a fellowship-trained rhinologist to ensure that the sinonasal cavity is otherwise healthy.

Subjects will be entered into the study in groups of three. The study will continue with successive cohorts of 3 subjects until dose-limiting toxicities (DLT) are observed in greater than 33% of the enrolled subjects. While escalating doses, we will monitor for signs or symptoms of toxicity. For the purposes of this trial, DLT will be defined as the development of statin intolerance with liver toxicity or muscle toxicity (as determined by elevated AST, ALT, or CK) or the development of significant systemic or sinonasal symptoms requiring drug discontinuation. We hypothesize that there will be no more than minimal side effects. Each participant will complete bloodwork (serum CK, AST, ALT) again at the completion of the study.

Weekly throughout the study, subjects will complete the Sino-Nasal Outcome Test-22 (SNOT-22, ©2006, Washington University, St. Louis, MO), a validated, patient-reported measure of sinonasal symptoms. The SNOT-22 evaluates physical, functional, and emotional consequences of sinonasal pathology using a Likert scale: 0= "None"; 1="Very mild"; 2="Mild or slight"; 3="Moderate"; 4="Severe"; and 5="As bad as it can be." The absolute change in SNOT-22 scores from baseline will be utilized to describe any adverse effects of simvastatin rinses on sinonasal function and quality of life.

Nasal endoscopy will also be performed by a fellowship-trained rhinologist within 6 months of study enrollment and at study completion to ensure no local tissue effects of topical simvastatin rinses. A Lund-Kennedy score, which reflect sinonasal disease severity, will be noted at the time of nasal endoscopy.

Olfactory function for each participant will also be evaluated at the time of initiation and completion of this study via the University of Pennsylvania Smell Identification Test (UPSIT). The UPSIT is a validated evaluation of olfaction acuity. Subjects smell 40 scratch-and-sniff items and then select the perceived odor in a choice manner from 4 scent options. Each correct smell identification is given a score of 1, resulting in final test scores of 1-40. Scores > 34 for males and > 35 for females are representative of normosmia. Score changes > 4 are considered clinically significant.

The current study would provide the support for Phase II and III clinical trials. Additionally, the study has applications for other disease processes affecting the sinonasal cavities.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-70 years old
2. Diagnosis of COVID-19 at least 3 months prior to study enrollment, but no greater than 12 months prior to study.
3. Objective olfactory dysfunction, believed to be due to COVID-19, that has persisted despite viral recovery otherwise (initial score on the UPSIT consistent with decreased olfactory function (<= 34 in women, <=33 in men)
4. Not currently using concomitant therapies specifically for the treamtment of OD, or willing to discontinue other therapies for the treatment of OD for the duration of the trial
5. Ability to read, write, and understand English

Exclusion Criteria:

1. Olfactory loss prior to COVID-19 infection
2. History of conditions that impact olfactory function

   1. Chronic rhinosinusitis
   2. History of prior sinonasal or skullbase surgery
   3. Neurodegenerative disorders (Parkinson's disease, Huntington's disease, Amyotrophic lateral sclerosis, Lewy body dementia, frontotemporal dementia)
3. Current or recent (within 8 weeks of study enrollment) oral statin use
4. History of conditions that increase risks of statin intolerance

   1. Untreated hypothyroidism
   2. History of chronic kidney disease or abnormal renal function at the time of enrollment
   3. Personal or family history of myositis or elevated creatine kinase at the time of enrollment
   4. Alcohol consumption greater than 7 drinks per week (female) or 14 drinks per week (male)
   5. History of liver disease or elevated liver enzymes at the time of enrollment
   6. History of statin intolerance
   7. Human immunodeficiency virus
   8. Viral hepatitis
5. History indicating that the subject should receive oral statins

   1. Angina
   2. Myocardialinfarction
   3. Cardiac surgery in the last 2 years
   4. Elevated total cholesterol at baseline
6. History of malignancy
7. History of statin intolerance
8. Currently pregnant or nursing
9. Use of any medications contraindicated with statins

   1. Antiviral protease inhibitors
   2. Macrolides
   3. Antifungals
   4. Cyclosporine
   5. Calcium channel blockers
   6. Diltiazem
   7. Danazole
   8. Amiodarone
   9. Gemfibrozil
   10. Nefazodone
   11. Ingestion of >1 quart of grapefruit juice per day
   12. Digoxin
   13. Niacin
   14. Coumadin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of simvastatin nasal wash | 4 weeks
  Primary objective is to evaluate safety and feasibility of simvastatin nasal wash.
  * Successive cohorts of 3 subjects will be enrolled until dose-limiting toxicities (DLT; defined as the development of statin intolerance with liver toxivity or muscle toxicity as determined by elevated AST, ALT, or CK or the development of significant systemic or sinonasal symptoms requiring drug discontinuation) are observed in greater than 33% of the enrolled subjects. We will monitor for signs or symptoms of toxicity.
  * Weekly throughout the study, subjects will complete the SNOT-22. The absolute change in SNOT-22 scores from baseline will be utilized to describe any adverse effects of simvastatin rinses on sinonasal function and quality of life.
  * Nasal endoscopy will be performed at the time of enrollment and at study completion to ensure no local tissue effects of topical simvastatin rinses. A Lund-Kennedy score reflecting sinonasal disease severity will be noted at the time of nasal endoscopy.

SECONDARY OUTCOMES:
Maximum tolerable dose of simvastatin nasal rinses via a dose escalation trial. | 4 weeks
  The secondary goal of this study is to determine the maximum tolerable dose of simvastatin nasal rinses via a dose-escalation trial. The first cohort will receive the lowest dose of simvastatin (0.1 mg) via nasal irrigation for 4 weeks. If none of the 3 subjects report toxicity, the next group of 3 subjects enrolled will receive the consecutive higher dose of simvastatin for 1 month to a maximum dose of (1mg). We plan to test the following doses: 0.1 mg, 0.25 mg, 0.5 mg, 1 mg.
  Subjects will complete the SNOT-22 weekly. The absolute change in SNOT-22 scores from baseline will be utilized to describe any adverse effects of simvastatin rinses on sinonasal function and quality of life.
  Nasal endoscopy will be performed within 6 months of enrollment and at study completion to ensure no local tissue effects of topical simvastatin rinses. A Lund-Kennedy score, which reflect sinonasal disease severity, will be noted at the time of nasal endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Nyssa F Farrell, MD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No